CLINICAL TRIAL: NCT02679040
Title: Histological Response Rate After Mastectomy and Immediate Breast Reconstruction at the End of Neoadjuvant Chemotherapy and Radiotherapy
Acronym: HIST-RIC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIST-RIC-IPC 2014-014
Record Dates: First submitted 2016-01-25; First posted 2016-02-10 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Drug Therapy; Anthracyclines; Docetaxel; Trastuzumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Immediate Mammary Reconstruction (Experimental): Chemotherapy, radiation therapy, mastectomy with immediate mammary reconstruction
  Interventions: Procedure: Immediate mammary reconstruction; Drug: Chemotherapy; Radiation: Radiation therapy

INTERVENTIONS:
Procedure: Immediate mammary reconstruction — Chemotherapy administration then radiotherapy and then surgery : mastectomy and immediate mammary reconstruction.
Drug: Chemotherapy — Chemotherapy treatment
  Other Names: anthracyclines and taxotere with or without Herceptin
Radiation: Radiation therapy — Radiation therapy

SUMMARY:
At present, it is widely admitted not proposing immediate mammary reconstruction when an adjuvant radiotherapy is indicated because of the significant change of the cosmetic result (profit) and it whatever is the technique of reconstruction adopted. This is true all the more as it is about a reconstruction by prosthesis because of the prothetic died risk of hull(shell).

Teams proposed immediate mammary reconstructions to expanding (carrier) patients of carcinoma infiltrating, sometimes locally moved forward. For these patients, was not brought back(reported) by increase of the risk of local or remote relapse.

Two studies estimated afterward the feasibility of the mastectomy with immediate mammary reconstruction at the close of the chemotherapy and of the radiotherapy. The rate of morbidity is judged as acceptable. The rate of local second offense(recurrence) was similar to the patients benefiting from the classic therapeutic plan.

During an other study ( M-RIC), it was shown that the inversion of therapeutic sequence is possible and that by prescribing the chemotherapy and the radiotherapy before immediate mammary reconstruction, the morbidity is acceptable.

It is acquired that the chemotherapy néoadjuvant is equivalent to the post-operative chemotherapy as regards the global survival.

On the other hand, the rate of histological answer, according to subgroups, is very different. This rate can vary of 9 % for tumors RH +, negative Her2 in 45 % for tumors RH-, Her2 over expression. There are 33 % for the RH +, Her2 + and of 35 % for triple-negative.

The purpose of the investigators study is to estimate the rate of histological response during the inversion of therapeutic sequence to make sure of the oncologic safety(security), in particular by molecular subgroups, considering the heterogeneousness of the results(profits) after chemotherapy néoadjuvant only. Sataloff and Chevallier Classifications is the references and will be used here, but the investigators can also use Symmans classification in addition.

The rate of local and metastatic second offenses(recurrences) will also be estimated.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years,
* Infiltrating carcinoma,
* Neoadjuvant chemotherapy indication,
* Radiotherapy indication,
* 0 or 1 score Performance status (WHO),
* Signed informed consent,
* Affiliation to Social Security System

Exclusion Criteria:

* Lobular carcinoma,
* "Luminal A" Tumor (RH+ and Her2 negative with grade I, and tumor RH+ Her2 negative with grade II and with Ki67<20%),
* Attempt of first conservative treatment,
* Metastatic breast cancer,
* Inflammatory carcinoma,
* History of homolateral or controlateral mammary carcinoma,
* Progression disease (despite neoadjuvant chemotherapy),
* Contraindications in an immediate mammary reconstruction by scrap of big dorsal (comorbidity),
* Any psychological, familial, sociological or geographical condition-potentially hampering compliance with the study protocol or follow-up schedule,
* Patients deprived of liberty or placed under the authority of a tutor.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2016-01-27 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Rate of histological response of an infiltrating tumor within various molecular subgroups | from surgery up to 1 month
  Tumor Histological response (group RH+ Her2+, group RH+ Her2-, group RH- Her2+, and group RH- Her2-)

SECONDARY OUTCOMES:
Rate of ganglionar response on the axillary lymph nodes after chemotherapy and radiotherapy néoadjuvant | from surgery up to 1 month
  Number of lymph nodes collected and number of positive lymph nodes

OTHER OUTCOMES:
Rate of local and metastatic relapse | from surgery up to 5 years
  Local and metastatic relapse evaluated by radiological exams (Echo-mammography and MRI)
Quality of life in post-operative at 4 months and at 1 year and patient satisfaction | Before surgery, at day 21, at 6 months and at 12 months
  Quality of life evaluated by questionnaire QLQ-C30
Rate of post-operative complications | from surgery up to 1 month
  Post operative complications evaluated by clinical exam
Quality of life in post-operative at 4 months and at 1 year and patient satisfaction | Before surgery, at day 21, at 6 months and at 12 months
  Quality of life evaluated by questionnaire QLQ-BR23
Quality of life in post-operative at 4 months and at 1 year and patient satisfaction | Before surgery, at day 21, at 6 months and at 12 months
  Quality of life evaluated by questionnaire BREAST-Qtm satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: BANNIER Marie, MD, PhD, Principal Investigator — Institut Paoli-Calmettes
Locations (10):
- France (10):
  - Institut Paoli-Calmettes, Marseille, Bouches-du-Rhône
  - Institut Paul Papin, Angers
  - Polyclinique Urbain V, Avignon
  - Capio-Clinique Belharra, Bayonne
  - Institut Bergonie, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Institut Oscar Lambret, Lille
  - Clinique Clementville, Montpellier
  - Icm - Institut Regional Du Cancer de Montpellier, Montpellier
  - Institut Jean Godinot, Reims

REFERENCES:
- See also: Institut paoli-calmettes — http://institutpaolicalmettes.fr